CLINICAL TRIAL: NCT02494232
Title: To Review the Management and Follow-up of Patients With Minor Thoracic Injuries Treated by Emergency Physicians.
Brief Title: Emergency Management of Minor Blunt Thoracic Trauma
Status: Completed | Type: Observational
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, faruk güngör, MD, Antalya Training and Research Hospital
Other Study IDs: antalya TRH
Record Dates: First submitted 2015-07-05; First posted 2015-07-10 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Thoracic Injuries,
Keywords: minor blunt thoracic trauma; physical examination
MeSH Terms: conditions — Thoracic Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- minor blunt thoracic trauma patient: demographic data, physical examination findings

SUMMARY:
Thoracic traumas are frequent causes of emergency department admissions and the third most common cause of death from trauma. Although emergency management of major thoracic traumas that have high mortality and morbidity were discussed and well-understood in detail in the literature, there are limited information regarding diagnosis, emergency management, treatment and follow-up after discharge of patients with minor blunt thoracic traumas.

The investigators aimed to investigate demographic data, physical examination findings, and the relationship between lung injury, emergency department final diagnosis, hospitalization, discharge and re-admission rates, effects of prescribed analgesics on pain and re-admissions of patients with a pre-diagnosis of minor blunt thoracic trauma on first admission.

ELIGIBILITY:
Inclusion Criteria:

* Glasgow Coma Scale (GCS) of 15
* stable vital signs
* admitted within the first 6 hours after injury

Exclusion Criteria:

* urgent and urgent triage category

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who admitted within the first 6 hours after injury to hospital due to blunt thoracic trauma without concomitant major injury were considered to have minor thoracic trauma and were included in the study
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2013-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
The incidence of lung injuries caused by minor thoracic traumas will be assessed by using questionnaire. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: faruk güngör, md, Study Chair — Antalya Education and Research Hospital, Department of Emergency Medicine
Locations (1):
- Antalya Training and Research Hospital, Department of Emergency, Antalya, Turkey (Türkiye)

REFERENCES:
- [Result] Shields JF, Emond M, Guimont C, Pigeon D. Acute minor thoracic injuries: evaluation of practice and follow-up in the emergency department. Can Fam Physician. 2010 Mar;56(3):e117-24. PMID 20228291